CLINICAL TRIAL: NCT01917162
Title: Multi-Center Clinical Evaluation of Two Daily Disposable Contact Lenses
Brief Title: Multi-Center Clinical Evaluation of Two Daily Disposable Contact Lenses (Study 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-13-033
Record Dates: First submitted 2013-08-04; First posted 2013-08-06 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Refractive Error
Keywords: contact lenses; daily disposable contact lenses; silicone hydrogel; contact lens comfort; near-sighted
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nelfilcon A/UltraFilcon B (Other): Nelfilcon A contact lenses, followed by UltraFilcon B contact lenses. Each product worn bilaterally for one week in a daily wear, daily disposable modality.
  Interventions: Device: Nelfilcon A contact lens; Device: UltraFilcon B contact lens
- UltraFilcon B/Nelfilcon A (Other): UltraFilcon B contact lenses, followed by Nelfilcon A contact lenses. Each product worn bilaterally for one week in a daily wear, daily disposable modality.
  Interventions: Device: Nelfilcon A contact lens; Device: UltraFilcon B contact lens

INTERVENTIONS:
Device: Nelfilcon A contact lens — Soft contact lens CE-marked for daily disposable wear.
  Other Names: DAILIES® AquaComfort Plus®
Device: UltraFilcon B contact lens — Silicone hydrogel soft contact lens CE-marked for daily disposable wear. Private-label versions may be used.
  Other Names: Procornea BYO Air Daily

SUMMARY:
The purpose of this study is to compare the subjective performance of two daily disposable contact lenses with respect to comfort and handling.

ELIGIBILITY:
Inclusion Criteria:

* Adapted soft contact lens wearer;
* Spherical distance contact lens prescription between -1.00 and -6.00 diopter (inclusive);
* Spectacle cylinder ≤0.75 diopter in the least astigmatic eye, ≤1.00 diopter in the other;
* Correctable to 6/9 (20/30) in both eyes;
* Read, understand, and sign the informed consent;
* Willing to comply with the wear schedule;
* Willing to comply with the study visit schedule;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any active corneal infection, injury or inflammation;
* Systemic or ocular allergies which might interfere with contact lens wear;
* Systemic or ocular disease which might interfere with contact lens wear;
* Strabismus or amblyopia;
* Corneal refractive surgery and any anterior segment surgery;
* Use of systemic/topical medication contraindicating contact lens wear;
* Use of gas permeable contact lenses within 1 month preceding the study;
* Participation in any concurrent clinical trial or in the last 30 days;
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Initial comfort | Baseline
  Initial Comfort (within 10-15 minutes of lens insertion) will be assessed bilaterally by the participant at time of dispense. Initial Comfort will be graded on a 1-10 scale (10=cannot be felt, 1=painful).

SECONDARY OUTCOMES:
End of Day Comfort | Day 7
  End of Day Comfort will be assessed by the participant as a retrospective, bilateral evaluation of 1 week of wear. End of Day Comfort will be graded on a 1-10 scale (10=cannot be felt, 1=painful).
Overall Comfort | Day 7
  Overall Comfort will be assessed by the participant as a retrospective, bilateral evaluation of 1 week of wear. Overall Comfort will be graded on a 1-10 scale (10=cannot be felt, 1=painful).
Overall Handling at Time of Removal | Day 7
  Overall Handling at Time of Removal will be assessed by the participant as a retrospective, bilateral evaluation of 1 week of wear. Overall Handling at Time of Removal will be graded on a 1-10 scale (10=excellent, very easy; 1=unmanageable).

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nick, Dipl. Ing., Study Director — Alcon Research
Locations (1):
- Visioncare Research Ltd, Farnham, Surrey, United Kingdom